CLINICAL TRIAL: NCT06772701
Title: Validation of the French Version of the Edinburgh Postnatal Depression Scale (EPDS) Postnatally in the Father
Acronym: EPDS-PERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2024-A00242-45
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Fathers included at the maternity hospital or through the mother take the Mini International Neuropsychiatric Interview and complete the PH-Q9, EPDS and socio-demographic questionnaires. Fathers included through the awareness campaign have only the PH-Q9, EPDS and socio-demographic questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fathers included at the maternity hospital or through their wife (Active Comparator): At inclusion, fathers included at the maternity hospital or through their wife take the Mini International Neuropsychiatric Interview and complete the EPDS book (PH-Q9, EPDS and socio-demographic questionnaire). 6 to 8 weeks after the birth of their child, they complete only EPDS book.
  Interventions: Diagnostic Test: Mini International Neuropsychiatric Interview; Other: EPDS book
- fathers includes through the awareness campaign (Experimental): At inclusion, fathers included through the awareness campaign have only the EPDS book (PH-Q9, EPDS and socio-demographic questionnaire) at inclusion. 6 to 8 weeks after the birth of their child, they complete the same EPDS book.
  Interventions: Other: EPDS book

INTERVENTIONS:
Diagnostic Test: Mini International Neuropsychiatric Interview — Fathers have Mini International Neuropsychiatric Interview, the standard diagnostic tool for post-natal depression
  Arms: Fathers included at the maternity hospital or through their wife
Other: EPDS book — PH-Q9, EPDS and socio-demographic questionnaires are completed online at inclusion and 6 to 8 weeks after the birth of child.

SUMMARY:
In recent years, fatherhood has changed considerably. Fathers are now more involved during the perinatal period, with their partner but also in caring for the child. Investigators now know that this period is also a source of major psychological upheaval, identity crisis, apprehension and anxiety for men. These upheavals can lead to depression that must be detected and treated as early as possible. This is an easy screening to perform using the EPDS (Edinburgh Postnatal Depression Scale). Currently, the EPDS is the most widely used self-questionnaire to assess the risk of depression in women during the perinatal period. Indeed, it is systematically recommended in many countries. It is starting to be used for the same purpose in the perinatal period in men, although the scale has not been validated in a representative sample of men in the pre- or post-natal period.

The main objective is to validate the use of the EPDS scale as a screening tool for postnatal depression in a population of French fathers.

They complete the PH-Q9, EPDS and socio-demographic questionnaires online at inclusion and 6 to 8 weeks after the birth of their child. Fathers included at the maternity ward also too Mini International Neuropsychiatric Interview (MINI) at inclusion.

DETAILED DESCRIPTION:
Fathers complete the PH-Q9, EPDS and socio-demographic questionnaires online at inclusion and 6 to 8 weeks after the birth of their child. Fathers included at the maternity ward also too Mini International Neuropsychiatric Interview (MINI) at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* All fathers whose baby is 10 days old or less

Exclusion Criteria:

* People with a poor understanding of spoken or written French
* Minors
* Persons under court protection, guardianship or curatorship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-03-12 (Estimated)

PRIMARY OUTCOMES:
Mini International Neuropsychiatric Interview | at inclusion
  This short structured clinical interview is used to diagnose psychiatric disorders and is currently the gold standard for diagnosing depression.

SECONDARY OUTCOMES:
socio-demographic questionnaire | at inclusion and 6 to 8 weeks after the birth of their child
  Socio-demographic data will be a secondary evaluation criterion. It will be used to study risk and protective factors, both those already known in the literature and those that have been little studied, and to identify profiles that are more at risk, with a view to taking preventive action in the field.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Antoine-Béclère hospital AP-HP, Clamart
  - Le Havre hospital - site Jacques Monod, Montivilliers

IPD SHARING:
Plan to Share IPD: No